CLINICAL TRIAL: NCT00578929
Title: Safety and Efficacy of Olopatadine HCl Nasal Spray in 6-11 Year Old Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Darrell Lange, Clinical Trial Manager, Alcon Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-07-01
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2010-02-09 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: allergic rhinitis; allergies; seasonal allergies
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Olopatadine 0.6% 1 Spray (Experimental): Olopatadine HCl 0.6% 1 spray per nostril twice daily
  Interventions: Drug: Olopatadine Hydrochloride Nasal Spray 0.6%
- Vehicle 1 spray (Placebo Comparator): Vehicle 1 spray per nostril twice daily
  Interventions: Drug: Vehicle
- Olopatadine 0.6% 2 sprays (Experimental): Olopatadine HCl 0.6% 2 sprays per nostril twice daily
  Interventions: Drug: Olopatadine Hydrochloride Nasal Spray 0.6%
- Vehicle 2 sprays (Placebo Comparator): Vehicle 2 sprays per nostril twice daily
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Olopatadine Hydrochloride Nasal Spray 0.6% — Olopatadine HCl 1 or 2 sprays per nostril twice daily
  Arms: Olopatadine 0.6% 1 Spray; Olopatadine 0.6% 2 sprays
Drug: Vehicle — Vehicle 1 or 2 sprays per nostril twice daily
  Arms: Vehicle 1 spray; Vehicle 2 sprays

SUMMARY:
A study to demonstrate the superiority of test article nasal spray relative to vehicle nasal spray for the treatment of seasonal allergic rhinitis for a 2 week period in patients aged 6 to 11 years with a history of seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; minimum of 6 years of age and less than 12 years
* 2 year history of seasonal allergic rhinitis

Exclusion Criteria:

* Concurrent disease that might interfere with the investigation or evaluation of te study medication
* Confirmed diagnosis of chronic rhinosinusitis within the last year
* Asthma, with the exception of mild intermittent asthma
* Anatomical nasal deformity
* Nasal obstruction
* Known non-responder to antihistamines for symptoms of Seasonal Allergic Rhinitis (SAR)
* Chronic or intermittent use of of inhaled, oral, intramuscular intravenous corticosteroids ot topical steroids
* Ocular disorder other that allergic conjunctivitis

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2388 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ed Tumaian, Study Director — ed.tumaian@alconlabs.com
Locations (1):
- Kenilworth/IL, Kenilworth, Illinois, United States

REFERENCES:
- [Derived] Meltzer EO, Blaiss M, Fairchild CJ. Comprehensive report of olopatadine 0.6% nasal spray as treatment for children with seasonal allergic rhinitis. Allergy Asthma Proc. 2011 May-Jun;32(3):213-20. doi: 10.2500/aap.2011.32.3448. Epub 2011 Apr 8. PMID 21477426

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled in the study on September 8, 2007 and the last subject exited the study on November 24, 2008. The study was conducted at medical clinics throughout the USA.
Pre-assignment Details: Subjects completed a 4-16 day run-in period on vehicle prior to randomization.
Period: Vehicle Run-In Period
Arm/Group | Olopatadine 0.6% 1 Spray | Vehicle 1 Spray | Olopatadine 0.6% 2 Sprays | Vehicle 2 Sprays
Started | 0 | 2388 | 0 | 0
Completed | 0 | 2388 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Randomized Period
Arm/Group | Olopatadine 0.6% 1 Spray | Vehicle 1 Spray | Olopatadine 0.6% 2 Sprays | Vehicle 2 Sprays
Started | 298 | 297 | 296 | 297
Completed | 281 | 283 | 288 | 283
Not Completed | 17 | 14 | 8 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olopatadine 0.6% 1 Spray | Vehicle 1 Spray | Olopatadine 0.6% 2 Sprays | Vehicle 2 Sprays | Total
Number analyzed (Participants) | 298 | 297 | 296 | 297 | 1188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 298 | 297 | 296 | 297 | 1188
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 125 | 122 | 124 | 501
  Male | 168 | 172 | 174 | 173 | 687

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Reflective Total Nasal Symptom Score (TNSS)
Description: Total Nasal Symptom Score comprised of scoring each of the following symptoms: runny nose, stuffy nose, itchy nose, and sneezing. Each symptom was scored as a 0 (none), 1 (mild), 2 (moderate), or 3 (severe). The 4 individual symptom scores were then added together for a total nasal symptom score.
  The percent change from baseline was defined as the average of the morning and evening severity scores for the sum of the assessments of the 4 individual scores averaged across all days.
Time Frame: Baseline through 2 weeks after randomization
Measure: Least Squares Mean (Standard Error); unit: Percent change of TNSS from baseline
Arm/Group | Olopatadine 0.6% 1 Spray | Vehicle 1 Spray | Olopatadine 0.6% 2 Sprays | Vehicle 2 Sprays
Number analyzed (Participants) | 298 | 297 | 296 | 297
Percent change of TNSS from baseline | -25.10 (1.45) | -18.17 (1.45) | -26.35 (1.45) | -21.21 (1.45)

2. Secondary Outcome: Percent Change From Baseline in the Reflective Total Ocular Symptom Score (TOSS)
Description: Total Ocular Symptom Score comprised of scoring each of the following symptoms: itchy eyes and watery eyes. Each symptom was scored as a 0 (none), 1 (mild), 2 (moderate), or 3 (severe). The 2 individual symptom scores were then added together for a total ocular symptom score.
  The percent change from baseline was defined as the average of the morning and evening severity scores for the sum of the assessments of the 2 individual scores averaged across all days.
Time Frame: Baseline through 2 weeks after randomization
Measure: Least Squares Mean (Standard Error); unit: Percent change of TOSS from baseline
Arm/Group | Olopatadine 0.6% 1 Spray | Vehicle 1 Spray | Olopatadine 0.6% 2 Sprays | Vehicle 2 Sprays
Number analyzed (Participants) | 298 | 297 | 296 | 297
Percent change of TOSS from baseline | -25.02 (5.11) | -6.09 (5.10) | -25.03 (3.33) | -9.46 (3.37)

ADVERSE EVENTS:
Time Frame: Up to 3 weeks
Description: Adverse events were collected from the time of first dose with vehicle run-in until study exit. Adverse events were both volunteered and solicited
Groups:
- Vehicle Run-in Period: Vehicle Run-in Period
Arm/Group | Olopatadine 0.6% 1 Spray | Vehicle 1 Spray | Olopatadine 0.6% 2 Sprays | Vehicle 2 Sprays | Vehicle Run-in Period
Serious Adverse Events (participants affected / at risk) | 0/298 | 0/297 | 0/296 | 0/297 | 1/2388
Other Adverse Events (participants affected / at risk) | 29/298 | 21/297 | 26/296 | 30/297 | 107/2388
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olopatadine 0.6% 1 Spray (N=298) | Vehicle 1 Spray (N=297) | Olopatadine 0.6% 2 Sprays (N=296) | Vehicle 2 Sprays (N=297) | Vehicle Run-in Period (N=2388)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olopatadine 0.6% 1 Spray (N=298) | Vehicle 1 Spray (N=297) | Olopatadine 0.6% 2 Sprays (N=296) | Vehicle 2 Sprays (N=297) | Vehicle Run-in Period (N=2388)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 11 (12) | 18 (19) | 16 (18) | 42 (44)
Headache (Nervous system disorders) | 13 (15) | 11 (11) | 9 (9) | 16 (16) | 68 (68)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right of review 60 days prior to any publication or presentation of information related to the study. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than study data and results. The Institution and the Primary Investigator agree not to publish any study related material other than above.